CLINICAL TRIAL: NCT04933331
Title: An Observational Multi-cite Study to Evaluate and Compare the Effectiveness of Various Tooth Specific Treatments in the Management of Early Caries Lesions
Brief Title: Early Caries Lesion Management Observational Study
Acronym: ELMO
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CareQuest Institute for Oral Health (Other)
Responsible Party: Principal Investigator, Laura Kibbe, Laura Kibbe, BSDH, Clinical Innovation Manager, CareQuest Institute for Oral Health
Other Study IDs: DQCI003
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Initial Caries; Arrested Dental Caries; Cavitated Caries; Dental Caries; Dental Caries in Children
Keywords: Curodont Repair Fluoride Plus; silver diamine fluoride; glass ionomer sealants; Fluoride Varnish; minimally invasive dentistry; non-invasive dentistry; Initial Caries; Arrested Dental Caries; dental caries; Cavitated Caries; Restorative Dental Treatment; Dental restorations
MeSH Terms: conditions — Dental Caries | interventions — Silver Staining; Sodium Fluoride; Clinpro Sealant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (4):
- Curodont Repair Fluoride Plus (Curodont) cohort: The effectiveness of Curodont treatment in this group will be compared to other treatment options and cohorts. Curodont will be professionally applied in the dental clinic. The treatment time takes about 5 minutes. Patients receive one professional dose application and be provided with homecare instructions and will be instructed to return for regular dental visits and exams according to the frequency determined by their dental team, usually every 6 months.
  Interventions: Drug: Curodont Repair Fluoride Plus; Device: Fluoride varnish; Drug: Fluoride toothpaste
- Other tooth-specific initial lesion interventional treatments cohort(s): Silver Diamine Fluoride (SDF). The treatment time is about 2 minutes.
  Glass Ionomer Sealants: The treatment time takes about 5 minutes per sealant. Typically four sealants are completed in one visit.
  All patients will be provided with homecare instructions and will be instructed to return for regular dental visits and exams according to the frequency determined by their dental team, usually every 6 months.
  Interventions: Device: Silver Diamine Fluoride; Device: Glass Ionomer Sealant; Device: Fluoride varnish; Drug: Fluoride toothpaste
- Control cohort, no tooth-specific treatment or whole mouth treatment.: If a patient or their caregivers choose no tooth-specific treatment, they will be included in the control cohort. This group includes patients who chose to receive no treatment at all, as well as those who choose whole mouth treatments such as: 2.26% fluoride varnish, 1.23% fluoride foam, and 5000 ppm fluoride prescription toothpaste.
  Interventions: Device: Fluoride varnish; Drug: Fluoride toothpaste
- Orthodontic cohort: Patients in active orthodontic care will be analyzed separately from other patients to account for the impact of orthodontic appliances on treatment outcomes. Orthodontic appliances are recognized by the American Dental Association Caries Risk Assessment as a risk factor for caries because they create dental plaque stagnation areas that are difficult to clean. Initial caries lesions are very frequently seen immediately surrounding orthodontic brackets (braces), yet continued plaque stagnation over the treated areas may heavily influence the success of any treatment. All groups/cohorts above will be represented in the orthodontic cohort in parallel.
  Interventions: Drug: Curodont Repair Fluoride Plus; Device: Silver Diamine Fluoride; Device: Glass Ionomer Sealant; Device: Fluoride varnish; Drug: Fluoride toothpaste

INTERVENTIONS:
Drug: Curodont Repair Fluoride Plus — Self-assembling peptide that integrates calcium and phosphate ions into the same hydroxyapatite that the enamel is made of through biomimetic re-mineralization. Amino acid sequence: CH3,COQQRFEWEFEQQ,NH2.
  Other Names: Curolox; p11-4
  Groups: Curodont Repair Fluoride Plus (Curodont) cohort; Orthodontic cohort
Device: Silver Diamine Fluoride — Silver diamine fluoride 38% is indicated for the treatment of dentinal hypersensitivity. SDF works by killing pathogenic organisms and hardens softened dentin making it more acid and abrasion resistant. The ADA recommends the use of SDF in treating early lesions.
  Other Names: SDF; Silver Nitrate
  Groups: Orthodontic cohort; Other tooth-specific initial lesion interventional treatments cohort(s)
Device: Glass Ionomer Sealant — A hydrophilic type of sealant material made with water, polymeric acid, and glass power. These sealants release fluoride over time which also helps protect against and repair initial caries lesions. The ADA recommends the use of sealants in treating occlusal early lesions.
  Other Names: GI Sealant
  Groups: Orthodontic cohort; Other tooth-specific initial lesion interventional treatments cohort(s)
Device: Fluoride varnish — 2.5% Sodium Fluoride Varnish which reduces dentinal hypersensitivity by occluding dentinal tubules.
Drug: Fluoride toothpaste — Prescription sodium fluoride toothpaste medicament used in place of regular toothpaste. It works by making the teeth stronger and more resistant to caries.
  Other Names: Prevident; Clinpro

SUMMARY:
The purpose of this observational study is to assess the effectiveness of Curodont Repair Fluoride Plus (CRFP) compared to other tooth-specific treatments (silver diamine fluoride (SDF), sealants, or other FDA-approved treatments) in preventing progression to cavitation in patients with at least one early non-cavitated dental caries lesion.

The study will also evaluate the effectiveness of CRFP in comparison to no tooth-specific treatment control groups, including whole mouth treatments such as: 2.26% fluoride varnish, 1.23% fluoride foam, and 5000 ppm fluoride prescription toothpaste; and no treatment, on caries arrest and in preventing progression to cavitation in patients with at least one early non-cavitated dental lesion.

DETAILED DESCRIPTION:
Study subjects will be enrolled upon diagnosis of at least one ADA Caries Classification system "initial" caries lesion. Subjects will be further sorted into study cohorts based on the non-invasive treatment option they select. The early lesions will be followed for 24 months after the date of the initial caries lesion diagnosis or the date of the first non-invasive treatment applied to the lesion.

Patients who choose CRFP will serve as the primary variable of interest. The primary objective is to assess the effectiveness of CRFP compared to other tooth specific treatments (SDF, sealants, or other FDA-approved treatments) in preventing progression to cavitation in initial dental lesions. The primary endpoint will be measured by the percentage of patients that require operative treatment for at least one early lesion noted at baseline during the following 24 months of observation.

The secondary objectives are to assess the effectiveness of CRFP compared to no tooth-specific treatment (including whole mouth treatments such as: fluoride varnish, fluoride foam, prescription toothpaste; other FDA-approved treatments; and no treatment) on 1.) caries arrest and 2.) preventing progression to cavitation in patients with at least one early dental lesion. The secondary endpoints will be measured by 1.) the percentage of patients that have caries arrest for at least one early lesion noted at baseline during the following 24 months of observation and 2.) the percentage of patients that require operative treatment for at least one early lesion noted at baseline during the following 24 months of observation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with permanent teeth who are diagnosed with at least one American Dental Association Caries Classification System (ADACCS) "Initial" caries lesion in a permanent tooth, will be included in this analysis.

Exclusion Criteria:

* Primary teeth
* Permanent teeth with ADACCS "Moderate" or "Advanced" caries lesions
* Healthy/ ADACCS "Sound" teeth

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This project will include patients of specified DentaQuest CareGroup clinics in Massachusetts, Alabama, Texas, and Oregon. There will be no special inclusion/exclusion criteria by race and/or ethnic origin.
  * The pediatric cohort will include patients with permanent teeth up to the 21st birthday.
  * The orthodontic cohort will include all ages.
  * The adult cohort will include all patients age 21 and above.
Sampling Method: Non-Probability Sample
Enrollment: 744 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
To assess the effectiveness of CRFP compared to other tooth specific treatments in preventing progression to cavitation. | 24 months
  The percentage of patients treated with CRFP that require operative treatment for at least one early lesion within the 24 months.

SECONDARY OUTCOMES:
To assess the effectiveness of CRFP compared to no tooth specific treatments (including whole mouth treatments) on caries arrest. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of patients that have caries arrest for at least one early lesion noted at baseline during the 24 months of observation from baseline.
To assess the effectiveness of CRFP compared to no tooth specific treatment (including whole mouth treatment) in preventing progression to cavitation. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of patients that require operative treatment for at least one early lesion noted at baseline during the 24 months of observation from baseline.

OTHER OUTCOMES:
To assess the effectiveness of SDF compared to no tooth specific treatment (including whole mouth treatment) on caries arrest in patients with at least one early dental lesion. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with SDF that have caries arrest for at least one early lesion noted at baseline during the 24 months of observation from baseline.
To assess the effectiveness of SDF (silver diamine fluoride) compared to no tooth specific treatment (including whole mouth treatment) in preventing progression to cavitation. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with SDF that require operative treatment for at least one early lesion noted at baseline during the 24 months of observation from baseline.
To assess the effectiveness of sealants compared to no tooth specific treatment (including whole mouth treatment) in preventing progression to cavitation. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with sealants that require operative treatment for at least one early lesion noted at baseline during the 24 months of observation from baseline.
To assess the effectiveness of CRFP compared to sealants in preventing progression to cavitation. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with CRFP that require operative treatment compared to those treated with sealants during the 24 months of observation from baseline.
To assess the effectiveness of CRFP compared to SDF in preventing progression to cavitation. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with CRFP that require operative treatment compared to those treated with SDF during the 24 months of observation from baseline.
To assess the effectiveness of CRFP compared to SDF (silver diamine fluoride) on caries arrest in patients with at least one early dental lesion. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with CRFP that have caries arrest compared to those treated with SDF that have caries arrest during the 24 months of observation from baseline.
To assess the effectiveness of sealants compared to SDF (silver diamine fluoride) in preventing progression to cavitation in patients with at least one early dental lesion. | Baseline, 6 months, 12 months, 18 months, 24 months
  The percentage of lesions treated with SDF that require operative treatment compared to those treated with sealants during the 24 months of observation from baseline.
To assess the effectiveness of tooth specific treatments in patients who are actively undergoing orthodontic care and have at least one early dental lesion. | Baseline, 6 months, 12 months, 18 months, 24 months
  A comparison of lesions that have caries arrest or require operative treatment for early lesion interventions during the 24 months of observation from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Laura J Skaret, BS, Principal Investigator — CareQuest Innovation Partners
Locations (4):
- United States (4):
  - Sarrell Dental Clinic, Dothan, Alabama
  - DentaQuest (Advantage Dental) Oral Health Center, Westborough, Massachusetts
  - Advantage Dental Oral Health Center, Bend, Oregon
  - Community Dental Care, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No
Study data will be deidentified and stored on a secure server. There will be no plans to release individual participant data.

REFERENCES:
- [Background] Brantley CF, Bader JD, Shugars DA, Nesbit SP. Does the cycle of rerestoration lead to larger restorations? J Am Dent Assoc. 1995 Oct;126(10):1407-13. doi: 10.14219/jada.archive.1995.0052. PMID 7594013
- [Background] Fleming E, Afful J. Prevalence of Total and Untreated Dental Caries Among Youth: United States, 2015-2016. NCHS Data Brief. 2018 Apr;(307):1-8. PMID 29717975
- [Background] Seirawan H, Faust S, Mulligan R. The impact of oral health on the academic performance of disadvantaged children. Am J Public Health. 2012 Sep;102(9):1729-34. doi: 10.2105/AJPH.2011.300478. Epub 2012 Jul 19. PMID 22813093
- [Background] Jackson SL, Vann WF Jr, Kotch JB, Pahel BT, Lee JY. Impact of poor oral health on children's school attendance and performance. Am J Public Health. 2011 Oct;101(10):1900-6. doi: 10.2105/AJPH.2010.200915. Epub 2011 Feb 17. PMID 21330579
- [Background] Slayton RL, Urquhart O, Araujo MWB, Fontana M, Guzman-Armstrong S, Nascimento MM, Novy BB, Tinanoff N, Weyant RJ, Wolff MS, Young DA, Zero DT, Tampi MP, Pilcher L, Banfield L, Carrasco-Labra A. Evidence-based clinical practice guideline on nonrestorative treatments for carious lesions: A report from the American Dental Association. J Am Dent Assoc. 2018 Oct;149(10):837-849.e19. doi: 10.1016/j.adaj.2018.07.002. PMID 30261951
- [Background] Wright JT, Crall JJ, Fontana M, Gillette EJ, Novy BB, Dhar V, Donly K, Hewlett ER, Quinonez RB, Chaffin J, Crespin M, Iafolla T, Siegal MD, Tampi MP, Graham L, Estrich C, Carrasco-Labra A. Evidence-based clinical practice guideline for the use of pit-and-fissure sealants: A report of the American Dental Association and the American Academy of Pediatric Dentistry. J Am Dent Assoc. 2016 Aug;147(8):672-682.e12. doi: 10.1016/j.adaj.2016.06.001. PMID 27470525
- [Background] Gao SS, Zhao IS, Hiraishi N, Duangthip D, Mei ML, Lo ECM, Chu CH. Clinical Trials of Silver Diamine Fluoride in Arresting Caries among Children: A Systematic Review. JDR Clin Trans Res. 2016 Oct;1(3):201-210. doi: 10.1177/2380084416661474. Epub 2016 Aug 20. PMID 30931743
- [Background] Kind L, Stevanovic S, Wuttig S, Wimberger S, Hofer J, Muller B, Pieles U. Biomimetic Remineralization of Carious Lesions by Self-Assembling Peptide. J Dent Res. 2017 Jul;96(7):790-797. doi: 10.1177/0022034517698419. Epub 2017 Mar 27. PMID 28346861
- [Background] Saha S, Yang XB, Wijayathunga N, Harris S, Feichtinger GA, Davies RPW, Kirkham J. A biomimetic self-assembling peptide promotes bone regeneration in vivo: A rat cranial defect study. Bone. 2019 Oct;127:602-611. doi: 10.1016/j.bone.2019.06.020. Epub 2019 Jul 24. PMID 31351196
- [Background] Welk A, Ratzmann A, Reich M, Krey KF, Schwahn C. Effect of self-assembling peptide P11-4 on orthodontic treatment-induced carious lesions. Sci Rep. 2020 Apr 22;10(1):6819. doi: 10.1038/s41598-020-63633-0. PMID 32321955
- [Background] Broseler F, Tietmann C, Bommer C, Drechsel T, Heinzel-Gutenbrunner M, Jepsen S. Randomised clinical trial investigating self-assembling peptide P11-4 in the treatment of early caries. Clin Oral Investig. 2020 Jan;24(1):123-132. doi: 10.1007/s00784-019-02901-4. Epub 2019 Apr 29. PMID 31037343
- [Background] Doberdoli D, Bommer C, Begzati A, Haliti F, Heinzel-Gutenbrunner M, Juric H. Randomized Clinical Trial investigating Self-Assembling Peptide P11-4 for Treatment of Early Occlusal Caries. Sci Rep. 2020 Mar 6;10(1):4195. doi: 10.1038/s41598-020-60815-8. PMID 32144336
- [Background] Gozetici B, Ozturk-Bozkurt F, Toz-Akalin T. Comparative Evaluation of Resin Infiltration and Remineralisation of Noncavitated Smooth Surface Caries Lesions: 6-month Results. Oral Health Prev Dent. 2019;17(2):99-106. doi: 10.3290/j.ohpd.a42203. PMID 30874252
- [Background] Alkilzy M, Tarabaih A, Santamaria RM, Splieth CH. Self-assembling Peptide P11-4 and Fluoride for Regenerating Enamel. J Dent Res. 2018 Feb;97(2):148-154. doi: 10.1177/0022034517730531. Epub 2017 Sep 11. PMID 28892645
- [Background] Brunton PA, Davies RP, Burke JL, Smith A, Aggeli A, Brookes SJ, Kirkham J. Treatment of early caries lesions using biomimetic self-assembling peptides--a clinical safety trial. Br Dent J. 2013 Aug;215(4):E6. doi: 10.1038/sj.bdj.2013.741. PMID 23969679
- [Derived] Shah SV, Kibbe LJ, Heaton LJ, Desrosiers C, Wittenborn J, Filipova M, Zaydenman K, Keeper JH. Framework for fiscal impact analysis of managing initial caries lesions with noninvasive therapies. J Am Dent Assoc. 2023 Oct;154(10):897-909.e6. doi: 10.1016/j.adaj.2023.07.007. PMID 37770132